CLINICAL TRIAL: NCT05883137
Title: High-flow Nasal Oxygenation for Apnoeic Oxygenation With Optiflow Switch During Intubation of the Critically Ill Adult- a Prospective Before-and-after Study
Brief Title: High-flow Nasal Oxygenation for Apnoeic Oxygenation During Intubation of the Critically Ill
Acronym: HiPOXIC
Status: Recruiting | Type: Observational
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-0063201
Record Dates: First submitted 2023-05-11; First posted 2023-05-31 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2024-11

CONDITIONS: Critical Illness; Respiratory Failure; Multi Organ Failure; Hypoxia
Keywords: Apnoeic oxygenation; Airway management; Intensive care; Critical care
MeSH Terms: conditions — Critical Illness; Respiratory Insufficiency; Multiple Organ Failure; Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Tight facemask or NIV: Preoxygenation with tight fitting facemask or NIV (non-invasive ventilation) according to the paitents need before anaesthesia induction.
- High Flow Nasal Oxygen and Tight facemask/ NIV: Pre and peri-oxygenation with HFNO using Optiflow Switch in addition to tight fitting facemask or NIV (non-invasive ventilation).
  Interventions: Device: Optiflow Switch

INTERVENTIONS:
Device: Optiflow Switch — High flow nasal oxygen with the Optiflow Switch device
  Groups: High Flow Nasal Oxygen and Tight facemask/ NIV

SUMMARY:
Intubation in the intensive care unit is a standard procedure with a high risk of adverse events such as hypoxaemia and cardiovascular instability. However, it is demonstrated that HFNO (High Flow Nasal Oxygen) for pre and perioxygenation is feasible and, in many situations, prolongs the safe apnoeic period after anaesthesia induction. Previous data of the use of HFNO during intubation of the critically ill is conflicting.

With the new device Optiflow Switch, which allow its combination with NIV or tight facemask with perioxygenation, we aim to evaluate whether this could reduce intubation-related hypoxaemia and other adverse events.

The general purpose of this project is to compare the addition of Optiflow Switch for pre- and perioxygenation to traditional preoxygenation using a tight-fitting mask or NIV during intubation in adult intensive care patients in a prospective before-and-after study design.

DETAILED DESCRIPTION:
This study aims to investigate whether apnoeic oxygenation with Optiflow Switch during tracheal intubation of the critically ill may prevent severe hypoxaemic events. Critically ill patients requiring intubation in the intensive care unit will be preoxygenated with tight facemask/NIV and Optiflow Switch or only tight facemask/ NIV.

During a period of 6-12 months with an aim to include a minimum of 50 patients, patients will be preoxygenated according to routine practice, 100% oxygen via a tight-fitting mask or NIV. During the following 6-12 months, we will change the clinical routine to adding HFNO with Optiflow Switch. During this time, patients, without contraindications will be pre and perioxygenated with HFNO, Optiflow Switch 40-70 L/min, 100 % O2, in combination with a tight facemask or NIV.

Before preoxygenation, the need for and methods for oxygen delivery is noted. Baseline patient characteristics (age, BMI, comorbidities, smoking history, airway related data) and the reason for intensive care admission and intubation will be registered. Scores for physiological compromise and length of intensive care prior to intubation will be noted.

In both groups, the duration of preoxygenation and drugs for anaesthesia induction are chosen by the intensive care physician responsible. Blood gas analysis for arterial oxygen and carbon dioxide partial pressure will be analysed before and after intubation. Before, during and after intubation, vital parameters will be registered.

Intubation-related data and immediate complications such as arterial hypotension, severe cardiac arrhythmia, cardiac arrest, death, oesophageal intubation, regurgitation, or a need for a surgical airway will be noted. Later complications such as ventilator-associated pneumonia and mortality at day 28 as well as duration of mechanical ventilation, length of stay in ICU will be registered.

Patients with contraindications against HFNO and if the responsible anaesthetist is not comfortable using HFNO will be preoxygenated with a traditional facemask or NIV and included in the study group of traditional preoxygenation.

Data will also be collected from the intensive care patient chart regarding all intubations during the study period in order to find patients not included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult, ≥18 years old
* Intensive care patients that require tracheal intubation for any indication

Exclusion Criteria:

* Patients with skull or facial injuries where the application of nasal cannula is to be avoided, decided by the intensivist.
* Pregnancy
* Total nasal obstruction
* Deemed not suitable for any other reason than the aforementioned

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult critically ill patients requiring intubation in the intensive care unit at Karolinska University Hospital Solna, Sweden will be included.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Desaturation up until 5 minutes after intubation | 5 minutes post intubation
  Desaturation (below 90% SpO2 or >5 % if <90% after preoxygenation) up until 5 minutes after intubation in patients receiving standard preoxygenation or with the addition of perioxygenation with HFNO.

SECONDARY OUTCOMES:
Frequency of complications | 5 minutes
  Difference of frequency of complications (severe arrhythmias or hypotension, cardiac arrest, death) when using Optiflow Switch peri-oxygenation compared to traditional preoxygenation.
Change of intubation method | 5 minutes
  Difference in change of intubation method when using Optiflow Switch peri-oxygenation compared to traditional preoxygenation.
Intensive care length of stay | 30 days
  Difference in long-time intensive care outcome (length of stay, 30-day mortality, ventilator-induced pneumonia) when using Optiflow Switch peri-oxygenation compared to traditional preoxygenation.
ETCO2 in the first breath after intubation | 5 minutes
  Difference in ETCO2 in the first breath after intubation when using Optiflow Switch peri-oxygenation compared to traditional preoxygenation.
Duration of intubation | 5 minutes
  Difference in duration of intubation (from the start of laryngoscopy until ETCO2 is registered) when using Optiflow Switch peri-oxygenation compared to traditional preoxygenation.
Arterial oxygen and carbon dioxide levels after intubation | 30 minutes
  Difference in arterial oxygen and carbon dioxide levels after intubation when using Optiflow Switch peri-oxygenation compared to traditional preoxygenation.
Perceived intubation difficulties | 30 minutes
  Difference in graded (scale 1-5) perceived difficulty during intubation when using Optiflow Switch peri-oxygenation compared to traditional preoxygenation.
Number of intubation attempts | 30 minutes
  Difference in number of intubation attempts when using Optiflow Switch peri-oxygenation compared to traditional preoxygenation.
Number of oesophageal intubations | 30 minutes
  Difference in number of oesophageal intubations when using Optiflow Switch peri-oxygenation compared to traditional preoxygenation.
30-day mortality | 30 days
  Difference in 30-day mortality when using Optiflow Switch peri-oxygenation compared to traditional preoxygenation.
Perceived operator stress | 30 minutes
  Difference in perceived operator stress during intubation when using Optiflow Switch peri-oxygenation compared to traditional preoxygenation.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No